CLINICAL TRIAL: NCT06146842
Title: A Trial to Determine the Optimal Bupivacaine Dose for Initiation of Labor Epidural Pain Relief with a Lidocaine Test Dose
Brief Title: ED90 of Bupivacaine After Lidocaine Test Dose with DPE and EPL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lawrence Ching Tsen, Associate Professor in Anaesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023p003001
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: A Randomized Biased-Coin Sequential Allocation Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DPE Group (Active Comparator): Subjects will receive an epidural catheter via a dural puncture epidural technique.
  Interventions: Drug: Bupivacaine Hydrochloride
- EPL Group (Active Comparator): Subjects will receive an epidural catheter via a traditional epidural technique.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — Each subject will receive allocated dose of bupivacaine

SUMMARY:
The primary objective of our study is to use a biased coin up-down allocation methodology to estimate the dose of bupivacaine required after the lidocaine test dose to achieve initial effective comfort in 90% of patients (post test-dose ED90) via the epidural (DPE or EPL) technique in women undergoing labor induction or augmentation; the investigators hypothesize that the investigators will be able to determine the post test-dose ED90 of bupivacaine for each technique with adequate precision to inform the optimal doses to study in a subsequent randomized trial comparing the analgesic effects of DPE vs. EPL. The investigators also hypothesize that the post test-dose ED90 of bupivacaine is lower with a DPE technique than with a conventional epidural technique.

DETAILED DESCRIPTION:
The investigators will be conducting a randomized controlled trial with patients randomized into either an EPL or a DPE group. For the first subject in the DPE and EPL techniques, the initial dose of bupivacaine 25 mg will be used, with an endpoint being the achievement of an NRS < 3 at 30 min. Subsequent patients are administered bupivacaine doses determined by the response of the previous subject, as per the biased coin method. The subsequent up and down interval doses are bupivacaine 2.5 mg (1 mL) increments. Hence, if the first subject does not respond successfully, the dose for the second subject will be bupivacaine 27.5 mg. If the second subject does not respond successfully, the dose for the third subject will be bupivacaine 30 mg. By contrast, if a subject responds successfully, the bupivacaine dose will be decreased to 22.5 mg with a probability of 10% and maintained with a probability of 90% (ratio 1:9).

ELIGIBILITY:
Inclusion Criteria:

1. Parturient with no major co-morbidities
2. Singleton, vertex gestation at term (37-42 weeks)
3. Less than or equal to 5 cm dilation
4. Desire to receive epidural labor analgesia
5. Numerical Rating Scale greater than or equal to 5 (NRS 0-10, where 0 = no pain, and 10 = worst pain imaginable), at time of epidural labor analgesia request.

Exclusion Criteria:

1. Current or historical evidence of clinically significant disease or condition, including diseases of pregnancy (i.e., preeclampsia, gestational diabetes)
2. Any contraindication to the administration of an epidural technique (e.g., thrombocytopenia, antiplatelet meds).
3. History of hypersensitivity or idiosyncratic reaction to an amide local anesthetic agent
4. Evidence of anticipated fetal complications (i.e., fetal anomalies, IUGR (Intrauterine Growth Restriction), oligohydramnios, polyhydramnios)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
NRS <3 at 30 min | 30 minutes after time 0.
  Adequate analgesia is defined as NRS score less than 3 at 30 minutes after time 0.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No